CLINICAL TRIAL: NCT01423942
Title: Maturation of the Autonomic Nervous System in Prematures
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, wamir, MD, Rambam Health Care Campus
Other Study IDs: RMB-0215-11
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Analysis, Event History

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to try to evaluate the maturation of the autonomic nervous system in prematures.

DETAILED DESCRIPTION:
To evaluate the maturation of the autonomic nervous system in prematures by using heart rate variability analyses.

ELIGIBILITY:
Inclusion Criteria:

* All prematures

Ages: 1 Day to 100 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Prematures
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Herat rate variability (HRV) characteristics | 3 years
  It is well known that maturation of the autonomic nervous system can be detected by heart rate variability in children. The purpose of this study is to apply HRV characteristics in premature infants and try to evaluate if there are noticable changes in these parameters both in "healthy" and diseased premature infants longitudinally during their stay at the NICU. Outcome measures to be studied are very low frequency ( VLF), low-frequency ( LF), high frequency (HF) frequency bands in the power spectrum density (PSD) of HRV records.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Weissman, MD, Principal Investigator — RMC
Locations (1):
- RMC, Haifa, Israel